CLINICAL TRIAL: NCT02321176
Title: Pharmacokinetics of Trans-resveratrol Based Nutritional Supplement and Its Three Metabolites in Human Eyes and Blood
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Huazhong University of Science and Technology (Other)
Responsible Party: Principal Investigator, Xufang Sun, Pharmacokinetics of Trans-resveratrol Based Nutritional Supplement and Its three Metabolites in Human Eyes and Blood, Huazhong University of Science and Technology
Allocation: Not Applicable | Model: Single Group | Masking: Single
Other Study IDs: Sun2
Record Dates: First submitted 2014-06-07; First posted 2014-12-22 (Estimated); Last update posted 2014-12-22 (Estimated); Status verified 2014-12

CONDITIONS: Eye Disease
MeSH Terms: conditions — Eye Diseases | interventions — Resveratrol

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- pharmacokinetics,trans-resveratrol (Experimental): tissues from the eyes of the surgery of patients who received 1 Longevinex containing 100 mg of trans resveratrol active ingredient brand capsule for three days
  Interventions: Drug: trans-resveratrol

INTERVENTIONS:
Drug: trans-resveratrol — patients received 100mg Longevinex everyday,total of three days
  1 capsule daily for one day containing 100 mg of trans resveratrol active ingredient
  Other Names: LONGEVINEX

SUMMARY:
There is blood-eye barrier in eyes,but some oral medicines can enter in the tissues of eyes.

The primary objective of the study is to study the Pharmacokinetics of Trans-resveratrol and Its three Metabolites in Human Eyes and Blood

DETAILED DESCRIPTION:
This was a single-blind, randomised study investigating single oral dose of LONGEVINEX in two groups of about 20 Patients with rhegmatogenous retinal detachment retinal detachment（males and females).The subjects received 100mg LONGEVINEX everyday,a total of three days before surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with rhegmatogenous retinal detachment.
2. Male and female patients 18-60 years of age.
3. nonsmokers or who smoke<10 cigarettes/day.
4. BMI ranging from 19 to 30 kg/m^2 were eligible for the study.
5. Patients were considered to be healthy on the basis of electrocardiogram (ECG), and clinical laboratory safety tests (haematology, plasma biochemistry, urinalysis and hepatitis B, hepatitis C and HIV serology) performed at screening.
6. Women use measures to avoid conception during the study period (e.g. oral contraceptives, intrauterine devices [IUDs], and condoms).
7. Avoid ingesting grapefruit, grapefruit juice or other grapefruit juice containing products, and any herbal-based nutrient supplement or prescribed medications( grapefruit, cranberry, blueberry products, peanuts and peanut butter, grape and grape products, and red wine ) during the same period of time.
8. patients should abstain from alcohol-containing beverages at least two days prior to and during the study.

Exclusion Criteria:

1. Uncontrolled Blood pressure exceeding diastolic pressure of 100 mm Hg (sitting) during the screening period and uncontrolled diabetes mellitus
2. Participation in another simultaneous medical investigation or trial
3. Renal failure requiring dialysis or renal transplant or liver dysfunction History of other disease,or other findings giving reasonable suspicion of a disease or condition that contraindicates the use an investigational drug, might affect interpretation of the results of the study, or render the subject at high risk from treatment complications.5.IOP over 30 mmHg.
4. Any previous retinal laser photocoagulation to the study eye in treatment naive. Any previous intravitreal injection in study eye (triamcinolone or other) in treatment naive.
5. Any previous vitrectomy in study eye (posterior or anterior associated with vitreous loss in cataract surgery). Intracapsular cataract extraction (posterior capsule needs to be present).
6. Aphakia or absence of the posterior capsule in the study eye, Structural damage to the center of the macula in the study eye preexisting to CRVO likely to preclude improvement in visual acuity following the resolution of macular edema, including atrophy of the retinal pigment epithelium, subretinal fibrosis, laser scar(s).

   -

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2014-03; Primary Completion 2015-04 (Estimated); Study Completion 2015-04 (Estimated)

PRIMARY OUTCOMES:
Tmax | up to three days
  1 capsule containing 100 mg of trans resveratrol active ingredient daily for three days.Than detect the concentrations of the tissues from the eyes of the surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Sun Xufang, Study Director — Department of Ophthalmology,Tongji Hospital, Tongji Medical College, Huazhong University of science and Technology
Locations (1):
- Tongji Medical College of HUST, Wuhan, Hubei, China